CLINICAL TRIAL: NCT03531541
Title: Transcutaneous Electrical Nerve Stimulation and Cervical Joint Manipulation on Pressure Pain Threshold
Brief Title: Hypoalgesic Effect of Electrical Current and Cervical Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Jonathan Daniel Telles, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: U1111-1212-5389
Record Dates: First submitted 2018-04-24; First posted 2018-05-21 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Pain
Keywords: TENS; cervical manipulation; pressure pain
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated into 4 groups: (G1) active TENS and CJM, (G2) placebo TENS and CJM, (G3) placebo TENS and active CJM, (G4) active TENS and placebo CJM.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The blinding will be assessed by examiner 2 (responsible for administering TENS) asking the participants which TENS intervention they think they received, with 3 options for the answer: "active," "placebo" or "don't know". The same questions will be asked by examiner 2 for CJM. Next, examiner 3 (responsible for administering CJM) will receive the blinding outcome and have 3 options for the answer: "active," "placebo" or "don't know". Examiner 1 will receive the blinding outcome will be asked: "Which group does the patient belong to: active TENS and CJM, active TENS and placebo CJM, placebo TENS and active CJM or placebo TENS and CJM" Their responses to these questions will be recorded and used to measure the adequacy of participants and examiners
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- active TENS and CJM (Active Comparator): The active unit will be applied with the patient in a supine position at a high frequency of 100 Hz, and pulse duration of 100 µs. Strong but comfortable intensity as dictated by each subject will be applied for 20 minutes.
  After application of TENS The examiner 3, who is responsible for cervical joint manipulation, will enter the room and stand at the head of the patient. Using the middle phalanx of the second finger of one hand, the examiner will apply pressure laterally on the joint processes of C6 and C7 vertebrae; the examiner will cradle the patient's opposite side with the other hand and then perform an ipsilateral inclination towards the C6, C7 segments, followed by a contralateral rotation to the tissue barrier to perform a high-velocity low-amplitude manipulation (thrust).
  Interventions: Device: Application of TENS; Device: CJM
- placebos TENS and CJM (Placebo Comparator): The application of placebo TENS will be at a frequency of 100 Hz and pulse duration of 100 µs for 30 seconds. After the initial 30 seconds, the current amplitude will gradually decrease over 15 seconds until it reaches zero value.
  Placebo CJM will be performed using an identical position to the active manipulation, however, for only 15 seconds, as proposed by some authors that have used placebo group in their studies[42-44]. The examiner shall not exert tension in the joint capsule of the segment to ensure the placebo effect
  Interventions: Device: Placebo TENS; Device: Placebo CJM
- placebo TENS and active CJM (Active Comparator): The application of placebo TENS will be at a frequency of 100 Hz and pulse duration of 100 µs for 30 seconds. After the initial 30 seconds, the current amplitude will gradually decrease over 15 seconds until it reaches zero value.
  After application of placebo TENS The examiner 3, who is responsible for cervical joint manipulation, will enter the room and stand at the head of the patient. Using the middle phalanx of the second finger of one hand, the examiner will apply pressure laterally on the joint processes of C6 and C7 vertebrae; the examiner will cradle the patient's opposite side with the other hand and then perform an ipsilateral inclination towards the C6, C7 segments, followed by a contralateral rotation.
  Interventions: Device: CJM; Device: Placebo TENS
- active TENS and placebo CJM (Active Comparator): The active unit will be applied with the patient in a supine position at a high frequency of 100 Hz, and pulse duration of 100 µs. Strong but comfortable intensity as dictated by each subject will be applied for 20 minutes.
  After application of placebo TENS The examiner 3, who is responsible for cervical joint manipulation, will enter the room and stand at the head of the patient. Using the middle phalanx of the second finger of one hand, the examiner will apply pressure laterally on the joint processes of C6 and C7 vertebrae; the examiner will cradle the patient's opposite side with the other hand and then perform an ipsilateral inclination towards the C6, C7 segments, followed by a contralateral rotation.
  Interventions: Device: Application of TENS; Device: Placebo CJM

INTERVENTIONS:
Device: Application of TENS — The subject's skin will be cleaned with mild soap and water. Two square self-adhesive electrodes (5x5cm) will be placed 1 cm below the olecranon of the ulna and 10 cm above the radiocarpal joint of the dominant hand, maintaining the PPT measurement region between two electrodes. Two identical TENS units will be used: an active and a placebo (Neurodyn Portable TENS, IBRAMED). The active unit will be applied with the patient in a supine position at a high frequency of 100 Hz, and pulse duration of 100 µs. Strong but comfortable intensity as dictated by each subject will be applied for 20 minutes. Participants will be asked about the intensity of TENS every 5 minutes, and if the intensity has faded, the intensity will be increased again to a strong but comfortable level.
  Other Names: Transcutaneous Electrical Nerve Stimulation (TENS)
  Arms: active TENS and CJM; active TENS and placebo CJM
Device: CJM — The examiner 3, who is responsible for cervical joint manipulation, will enter the room and stand at the head of the patient. Using the middle phalanx of the second finger of one hand, the examiner will apply pressure laterally on the joint processes of C6 and C7 vertebrae; the examiner will cradle the patient's opposite side with the other hand and then perform an ipsilateral inclination towards the C6, C7 segments, followed by a contralateral rotation to the tissue barrier to perform a high-velocity low-amplitude manipulation (thrust). If the patient does not experience joint cavitation during the maneuver, two more attempts will be made. If no sound occurs on the third attempt, the joints will be considered manipulated.
  Other Names: Cervical Joint Manipulation
  Arms: active TENS and CJM; placebo TENS and active CJM
Device: Placebo TENS — The application of placebo TENS will be at a frequency of 100 Hz and pulse duration of 100 µs for 30 seconds. After the initial 30 seconds, the current amplitude will gradually decrease over 15 seconds until it reaches zero value. Participants will be informed that TENS can cause a slight tingling sensation or any sensation during the procedure. They will be asked every 5 minutes if they are comfortable, without increasing intensity as in the active TENS group
  Other Names: Placebo Transcutaneous Electrical Nerve Stimulation (TENS)
  Arms: placebo TENS and active CJM; placebos TENS and CJM
Device: Placebo CJM — Placebo CJM will be performed using an identical position to the active manipulation, however, for only 15 seconds, as proposed by some authors that have used placebo group in their studies. The examiner shall not exert tension in the joint capsule of the segment to ensure the placebo effect. The maneuvers will be carried out by a physiotherapist with more than 5 years of experience in manual therapy. The active or placebo manipulation will be performed on the right or left side according to randomization.
  Other Names: Placebo Cervical Joint Manipulation
  Arms: active TENS and placebo CJM; placebos TENS and CJM

SUMMARY:
This study evaluates the hypoalgesic effect of the TENS application associated with joint manipulation of the cervical region in healthy individuals. One group had both active treatments, the other group received both placebo treatments, the third and fourth group received only one of the two treatments actively and the other placebo

DETAILED DESCRIPTION:
Transcutaneous Electrical Nerve Stimulation (TENS) and Cervical Joint Manipulation (CJM) are often used for pain treatment.

TENS also promotes analgesia by activating a descending pathway, which originates in the periaqueductal grey (PAG) and in the rostroventromedial medulla (RVM) to inhibit the excitability of nociceptive neurons in the dorsal horn of the spinal cord.

Joint manipulation generates a series of stimuli within the central nervous system through the activation of proprioceptors located in the joint capsule or muscles, stimulates the PAG, causing pain inhibition by activation of non-opioid descending inhibitory pathways

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* no pain complaints from the last 90 days

Exclusion Criteria:

* previous spinal surgeries
* spinal canal stenosis
* vertebral fracture
* spondylolisthesis
* cancer
* acute infections
* hemorrhagic disorders
* active tuberculosis
* deep vein thrombosis
* osteoporosis
* diseases rheumatic
* diseases metabolic
* cardiorespiratory diseases
* headache in the last seven days
* smoking
* changes in skin sensitivity
* use of pacemaker
* women in menstrual period
* pregnant women
* use of pain-killers in the last 48 hours
* use of anti-inflammatory drugs in the last 48 hours
* previous electrostimulation
* previous cervical joint manipulation treatments
* hypersensitivity to TENS application
* aversion to cervical joint manipulation
* positive test for vertebral artery.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-01-27 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold of the posterior region of the forearm | 1 minute after the end of the intervention.
  The examiner will use a Somedic Type II digital pressure algometer (Somedic Inc, Hörby, Sweden) on the posterior region of the forearm 10cm below the lateral epicondyle of the elbow towards the third finger, with the forearm maintained in pronation. Next, the pressure will be applied perpendicularly to the skin at a rate of 40kPa/s using a flat, 1cm2 circular probe covered with 1mm of rubber to avoid any skin pain from sharp metal edges. The average of the PPT scores (in kPa) will be recorded by the assessor.

SECONDARY OUTCOMES:
Pressure Pain Threshold of the posterior region of the forearm | 20 minutes after the end of the intervention
  The examiner will use a Somedic Type II digital pressure algometer (Somedic Inc, Hörby, Sweden) on the posterior region of the forearm 10cm below the lateral epicondyle of the elbow towards the third finger, with the forearm maintained in pronation. Next, the pressure will be applied perpendicularly to the skin at a rate of 40kPa/s using a flat, 1cm2 circular probe covered with 1mm of rubber to avoid any skin pain from sharp metal edges. The average of the PPT scores (in kPa) will be recorded by the assessor.
Pressure Pain Threshold of the tibialis anterior muscle | 1 minute after the end of the intervention.
  For the PPT assessment over the tibialis anterior muscle of the dominant side, the patient will be positioned supine on a stretcher with the knees flexed at 90°. The examiner will place the pressure algometer 5 cm below the tibial tuberosity and 2.5 cm laterally to the tibial tuberosity over the tibialis anterior muscle.
Pressure Pain Threshold of the tibialis anterior muscle | 20 minutes after the end of the intervention
  For the PPT assessment over the tibialis anterior muscle of the dominant side, the patient will be positioned supine on a stretcher with the knees flexed at 90°. The examiner will place the pressure algometer 5 cm below the tibial tuberosity and 2.5 cm laterally to the tibial tuberosity over the tibialis anterior muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Liebano, Dr., Principal Investigator — Universidade Federal de São Carlos - UFScar
Locations (2):
- Brazil (2):
  - Centro Universitário Católico Salesiano Auxilium de Lins, Lins, São Paulo
  - Ufscar - Universidade Federal de São Carlos, São Carlos, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sluka KA, Deacon M, Stibal A, Strissel S, Terpstra A. Spinal blockade of opioid receptors prevents the analgesia produced by TENS in arthritic rats. J Pharmacol Exp Ther. 1999 May;289(2):840-6. PMID 10215661
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Mayer DJ, Price DD, Rafii A. Antagonism of acupuncture analgesia in man by the narcotic antagonist naloxone. Brain Res. 1977 Feb;121(2):368-72. doi: 10.1016/0006-8993(77)90161-5. No abstract available. PMID 832169
- [Background] Ha H, Tan EC, Fukunaga H, Aochi O. Naloxone reversal of acupuncture analgesia in the monkey. Exp Neurol. 1981 Jul;73(1):298-303. doi: 10.1016/0014-4886(81)90063-7. No abstract available. PMID 7250283
- [Background] Citak Karakaya I, Karakaya MG, Ergun E, Elmali S, Firat T. Effects of different frequencies of conventional transcutaneous electrical nerve stimulation on pressure pain threshold and tolerance. J Back Musculoskelet Rehabil. 2014;27(2):197-201. doi: 10.3233/BMR-130436. PMID 24254493
- [Background] Dailey DL, Rakel BA, Vance CGT, Liebano RE, Amrit AS, Bush HM, Lee KS, Lee JE, Sluka KA. Transcutaneous electrical nerve stimulation reduces pain, fatigue and hyperalgesia while restoring central inhibition in primary fibromyalgia. Pain. 2013 Nov;154(11):2554-2562. doi: 10.1016/j.pain.2013.07.043. Epub 2013 Jul 27. PMID 23900134
- [Background] Sabino GS, Santos CM, Francischi JN, de Resende MA. Release of endogenous opioids following transcutaneous electric nerve stimulation in an experimental model of acute inflammatory pain. J Pain. 2008 Feb;9(2):157-63. doi: 10.1016/j.jpain.2007.09.003. Epub 2007 Nov 7. PMID 17988952
- [Background] Chandran P, Sluka KA. Development of opioid tolerance with repeated transcutaneous electrical nerve stimulation administration. Pain. 2003 Mar;102(1-2):195-201. doi: 10.1016/s0304-3959(02)00381-0. PMID 12620611
- [Background] Han JS, Chen XH, Sun SL, Xu XJ, Yuan Y, Yan SC, Hao JX, Terenius L. Effect of low- and high-frequency TENS on Met-enkephalin-Arg-Phe and dynorphin A immunoreactivity in human lumbar CSF. Pain. 1991 Dec;47(3):295-298. doi: 10.1016/0304-3959(91)90218-M. PMID 1686080
- [Background] Flynn TW, Childs JD, Fritz JM. The audible pop from high-velocity thrust manipulation and outcome in individuals with low back pain. J Manipulative Physiol Ther. 2006 Jan;29(1):40-5. doi: 10.1016/j.jmpt.2005.11.005. PMID 16396728
- [Background] Dunning J, Rushton A. The effects of cervical high-velocity low-amplitude thrust manipulation on resting electromyographic activity of the biceps brachii muscle. Man Ther. 2009 Oct;14(5):508-13. doi: 10.1016/j.math.2008.09.003. Epub 2008 Nov 21. PMID 19027344
- [Background] DeVocht JW, Pickar JG, Wilder DG. Spinal manipulation alters electromyographic activity of paraspinal muscles: a descriptive study. J Manipulative Physiol Ther. 2005 Sep;28(7):465-71. doi: 10.1016/j.jmpt.2005.07.002. PMID 16182019
- [Background] Evans DW. Mechanisms and effects of spinal high-velocity, low-amplitude thrust manipulation: previous theories. J Manipulative Physiol Ther. 2002 May;25(4):251-62. doi: 10.1067/mmt.2002.123166. PMID 12021744
- [Background] Achalandabaso A, Plaza-Manzano G, Lomas-Vega R, Martinez-Amat A, Camacho MV, Gasso M, Hita-Contreras F, Molina F. Tissue damage markers after a spinal manipulation in healthy subjects: a preliminary report of a randomized controlled trial. Dis Markers. 2014;2014:815379. doi: 10.1155/2014/815379. Epub 2014 Dec 25. PMID 25609853
- [Background] Wright A. Hypoalgesia post-manipulative therapy: a review of a potential neurophysiological mechanism. Man Ther. 1995 Nov;1(1):11-6. doi: 10.1054/math.1995.0244. PMID 11327789
- [Background] Pickar JG, Wheeler JD. Response of muscle proprioceptors to spinal manipulative-like loads in the anesthetized cat. J Manipulative Physiol Ther. 2001 Jan;24(1):2-11. doi: 10.1067/mmt.2001.112017. PMID 11174689
- [Background] Maigne JY, Vautravers P. Mechanism of action of spinal manipulative therapy. Joint Bone Spine. 2003 Sep;70(5):336-41. doi: 10.1016/s1297-319x(03)00074-5. PMID 14563460
- [Background] Randoll C, Gagnon-Normandin V, Tessier J, Bois S, Rustamov N, O'Shaughnessy J, Descarreaux M, Piche M. The mechanism of back pain relief by spinal manipulation relies on decreased temporal summation of pain. Neuroscience. 2017 May 4;349:220-228. doi: 10.1016/j.neuroscience.2017.03.006. Epub 2017 Mar 11. PMID 28288900
- [Background] Bialosky JE, Bishop MD, Price DD, Robinson ME, George SZ. The mechanisms of manual therapy in the treatment of musculoskeletal pain: a comprehensive model. Man Ther. 2009 Oct;14(5):531-8. doi: 10.1016/j.math.2008.09.001. Epub 2008 Nov 21. PMID 19027342
- [Background] Coronado RA, Gay CW, Bialosky JE, Carnaby GD, Bishop MD, George SZ. Changes in pain sensitivity following spinal manipulation: a systematic review and meta-analysis. J Electromyogr Kinesiol. 2012 Oct;22(5):752-67. doi: 10.1016/j.jelekin.2011.12.013. Epub 2012 Jan 30. PMID 22296867
- [Background] Savva C, Giakas G, Efstathiou M. The role of the descending inhibitory pain mechanism in musculoskeletal pain following high-velocity, low amplitude thrust manipulation: a review of the literature. J Back Musculoskelet Rehabil. 2014;27(4):377-82. doi: 10.3233/BMR-140472. PMID 24867897
- [Background] Gay CW, Robinson ME, George SZ, Perlstein WM, Bishop MD. Immediate changes after manual therapy in resting-state functional connectivity as measured by functional magnetic resonance imaging in participants with induced low back pain. J Manipulative Physiol Ther. 2014 Nov-Dec;37(9):614-27. doi: 10.1016/j.jmpt.2014.09.001. Epub 2014 Oct 3. PMID 25284739
- [Background] Jordon MK, Beattie PF, D'Urso S, Scriven S. Spinal manipulation does not affect pressure pain thresholds in the absence of neuromodulators: a randomized controlled trial. J Man Manip Ther. 2017 Sep;25(4):172-181. doi: 10.1080/10669817.2016.1230352. Epub 2016 Sep 12. PMID 28912629
- [Background] Boal RW, Gillette RG. Central neuronal plasticity, low back pain and spinal manipulative therapy. J Manipulative Physiol Ther. 2004 Jun;27(5):314-26. doi: 10.1016/j.jmpt.2004.04.005. PMID 15195039
- [Background] Molina-Ortega F, Lomas-Vega R, Hita-Contreras F, Plaza Manzano G, Achalandabaso A, Ramos-Morcillo AJ, Martinez-Amat A. Immediate effects of spinal manipulation on nitric oxide, substance P and pain perception. Man Ther. 2014 Oct;19(5):411-7. doi: 10.1016/j.math.2014.02.007. Epub 2014 Mar 5. PMID 24674816
- [Background] Nakatsuka T, Chen M, Takeda D, King C, Ling J, Xing H, Ataka T, Vierck C, Yezierski R, Gu JG. Substance P-driven feed-forward inhibitory activity in the mammalian spinal cord. Mol Pain. 2005 Jun 29;1:20. doi: 10.1186/1744-8069-1-20. PMID 15987503
- [Background] Wu LJ, Xu H, Ko SW, Yoshimura M, Zhuo M. Feed-forward inhibition: a novel cellular mechanism for the analgesic effect of substance P. Mol Pain. 2005 Nov 18;1:34. doi: 10.1186/1744-8069-1-34. PMID 16297242
- [Background] Pantaleao MA, Laurino MF, Gallego NL, Cabral CM, Rakel B, Vance C, Sluka KA, Walsh DM, Liebano RE. Adjusting pulse amplitude during transcutaneous electrical nerve stimulation (TENS) application produces greater hypoalgesia. J Pain. 2011 May;12(5):581-90. doi: 10.1016/j.jpain.2010.11.001. Epub 2011 Feb 1. PMID 21277840
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Liebano RE, Rakel B, Vance CGT, Walsh DM, Sluka KA. An investigation of the development of analgesic tolerance to TENS in humans. Pain. 2011 Feb;152(2):335-342. doi: 10.1016/j.pain.2010.10.040. Epub 2010 Dec 8. PMID 21144659
- [Background] Leffler AS, Hansson P, Kosek E. Somatosensory perception in patients suffering from long-term trapezius myalgia at the site overlying the most painful part of the muscle and in an area of pain referral. Eur J Pain. 2003;7(3):267-76. doi: 10.1016/S1090-3801(02)00138-6. PMID 12725850
- [Background] Liebano RE, Vance CG, Rakel BA, Lee JE, Cooper NA, Marchand S, Walsh DM, Sluka KA. Transcutaneous electrical nerve stimulation and conditioned pain modulation influence the perception of pain in humans. Eur J Pain. 2013 Nov;17(10):1539-46. doi: 10.1002/j.1532-2149.2013.00328.x. Epub 2013 May 6. PMID 23650092
- [Background] Walton DM, Macdermid JC, Nielson W, Teasell RW, Chiasson M, Brown L. Reliability, standard error, and minimum detectable change of clinical pressure pain threshold testing in people with and without acute neck pain. J Orthop Sports Phys Ther. 2011 Sep;41(9):644-50. doi: 10.2519/jospt.2011.3666. Epub 2011 Sep 1. PMID 21885906
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Staud R. Treatment of fibromyalgia and its symptoms. Expert Opin Pharmacother. 2007 Aug;8(11):1629-42. doi: 10.1517/14656566.8.11.1629. PMID 17685881
- [Background] Moran F, Leonard T, Hawthorne S, Hughes CM, McCrum-Gardner E, Johnson MI, Rakel BA, Sluka KA, Walsh DM. Hypoalgesia in response to transcutaneous electrical nerve stimulation (TENS) depends on stimulation intensity. J Pain. 2011 Aug;12(8):929-35. doi: 10.1016/j.jpain.2011.02.352. Epub 2011 Apr 9. PMID 21481649
- [Background] Rakel B, Cooper N, Adams HJ, Messer BR, Frey Law LA, Dannen DR, Miller CA, Polehna AC, Ruggle RC, Vance CG, Walsh DM, Sluka KA. A new transient sham TENS device allows for investigator blinding while delivering a true placebo treatment. J Pain. 2010 Mar;11(3):230-8. doi: 10.1016/j.jpain.2009.07.007. Epub 2009 Nov 27. PMID 19945354
- [Background] Fernandez-Carnero J, Fernandez-de-Las-Penas C, de la Llave-Rincon AI, Ge HY, Arendt-Nielsen L. Widespread mechanical pain hypersensitivity as sign of central sensitization in unilateral epicondylalgia: a blinded, controlled study. Clin J Pain. 2009 Sep;25(7):555-61. doi: 10.1097/AJP.0b013e3181a68a040. PMID 19692795
- [Background] Saiz-Llamosas JR, Fernandez-Perez AM, Fajardo-Rodriguez MF, Pilat A, Valenza-Demet G, Fernandez-de-Las-Penas C. Changes in neck mobility and pressure pain threshold levels following a cervical myofascial induction technique in pain-free healthy subjects. J Manipulative Physiol Ther. 2009 Jun;32(5):352-7. doi: 10.1016/j.jmpt.2009.04.009. PMID 19539117
- [Background] Fernandez-de-las-Penas C, Perez-de-Heredia M, Brea-Rivero M, Miangolarra-Page JC. Immediate effects on pressure pain threshold following a single cervical spine manipulation in healthy subjects. J Orthop Sports Phys Ther. 2007 Jun;37(6):325-9. doi: 10.2519/jospt.2007.2542. PMID 17612359
- [Background] Vernon HT, Triano JJ, Ross JK, Tran SK, Soave DM, Dinulos MD. Validation of a novel sham cervical manipulation procedure. Spine J. 2012 Nov;12(11):1021-8. doi: 10.1016/j.spinee.2012.10.009. Epub 2012 Nov 15. PMID 23158966
- [Background] Gomes Ade O, Silvestre AC, Silva CF, Gomes MR, Bonfleur ML, Bertolini GR. Influence of different frequencies of transcutaneous electrical nerve stimulation on the threshold and pain intensity in young subjects. Einstein (Sao Paulo). 2014 Sep;12(3):318-22. doi: 10.1590/s1679-45082014ao3092. PMID 25295453
- [Background] Wassinger CA, Rich D, Cameron N, Clark S, Davenport S, Lingelbach M, Smith A, Baxter GD, Davidson J. Cervical & thoracic manipulations: Acute effects upon pain pressure threshold and self-reported pain in experimentally induced shoulder pain. Man Ther. 2016 Feb;21:227-32. doi: 10.1016/j.math.2015.08.009. Epub 2015 Aug 28. PMID 26391291
- [Background] Chesterton LS, Foster NE, Wright CC, Baxter GD, Barlas P. Effects of TENS frequency, intensity and stimulation site parameter manipulation on pressure pain thresholds in healthy human subjects. Pain. 2003 Nov;106(1-2):73-80. doi: 10.1016/s0304-3959(03)00292-6. PMID 14581113
- [Background] Tanaka K, Ikeuchi M, Izumi M, Aso K, Sugimura N, Enoki H, Nagano Y, Ishida K, Tani T. Effects of two different intensities of transcutaneous electrical nerve stimulation on pain thresholds of contralateral muscles in healthy subjects. J Phys Ther Sci. 2015 Sep;27(9):2771-4. doi: 10.1589/jpts.27.2771. Epub 2015 Sep 30. PMID 26504290
- [Background] Fernandez-Carnero J, Fernandez-de-las-Penas C, Cleland JA. Immediate hypoalgesic and motor effects after a single cervical spine manipulation in subjects with lateral epicondylalgia. J Manipulative Physiol Ther. 2008 Nov-Dec;31(9):675-81. doi: 10.1016/j.jmpt.2008.10.005. PMID 19028251
- [Result] Desantana JM, Sluka KA, Lauretti GR. High and low frequency TENS reduce postoperative pain intensity after laparoscopic tubal ligation: a randomized controlled trial. Clin J Pain. 2009 Jan;25(1):12-9. doi: 10.1097/AJP.0b013e31817d1070. PMID 19158541
- [Derived] Telles JD, Gabanela Schiavon MA, Rampazo da Silva EP, Liebano RE. Transcutaneous electrical nerve stimulation and cervical joint manipulation on pressure pain threshold. Pain Manag. 2018 Jul 1;8(4):263-269. doi: 10.2217/pmt-2017-0069. Epub 2018 Jun 1. PMID 29856269
- See also: The effect of manipulation and mobilisation on pressure pain thresholds in the thoracic spine — http://vuir.vu.edu.au/500/1/Manipulation_and_mobilisation_2004.pdf